CLINICAL TRIAL: NCT01057810
Title: Randomized, Double-Blind, Phase 3 Trial to Compare the Efficacy of Ipilimumab vs Placebo in Asymptomatic or Minimally Symptomatic Patients With Metastatic Chemotherapy-Naïve Castration Resistant Prostate Cancer
Brief Title: Phase 3 Study of Immunotherapy to Treat Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-095; 2009-016217-23 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab (Experimental)
  Interventions: Drug: Ipilimumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ipilimumab — 5 mg/ml solution, Intravenous, 10 mg/kg, Every 3 weeks for up to 4 doses in the Induction Phase. Every 12 weeks in the Maintenance Phase. Up to 24 weeks in the Induction Phase. Treatment in the Maintenance Phase continues until total treatment period has reached three years,Treatment Stopping Criteria are met, withdrawal of consent, or study closure
  Other Names: BMS-734016; MDX010
  Arms: Ipilimumab
Drug: Placebo — Solution, Intravenous, 0 mg, Every 3 weeks for up to 4 doses in the Induction Phase. Every 12 weeks in the Maintenance Phase. Up to 24 weeks in the Induction Phase. Treatment in the Maintenance Phase continues until total treatment period has reached three years,Treatment Stopping Criteria are met, withdrawal of consent, or study closure
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if asymptomatic or minimally symptomatic patients with metastatic prostate cancer who have not received chemotherapy live longer when treated with ipilimumab than those treated with a placebo

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Metastatic prostate cancer
* Asymptomatic or minimally symptomatic
* Progression during hormonal therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1

Exclusion Criteria:

* Liver, lung or brain metastases
* Prior immunotherapy or chemotherapy for metastatic prostate cancer
* Autoimmune disease
* HIV, Hepatitis B, or Hepatitis C infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2010-07; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (126):
- United States (42):
  - Alaska Clinical Research Center, Llc, Anchorage, Alaska
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Desert Hematology Oncology, Rancho Mirage, California
  - Southern California Permanente Medical Group, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - Lynn Cancer Institute Center For Hematology-Oncology, Boca Raton, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - Hematology Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida
  - Northside Hospital, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Gwinnett Hospital System Inc., Lawrenceville, Georgia
  - Straub Clinic And Hospital, Honolulu, Hawaii
  - University Of Chicago, Chicago, Illinois
  - Cancer Care Specialists Of Central Illinois, Decatur, Illinois
  - Goshen Center For Cancer Care, Goshen, Indiana
  - Hutchinson Clinic, Pa, Hutchinson, Kansas
  - Cancer Center Of Kansas, Wichita, Kansas
  - University Of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Goshen Medical Associates, Goshen, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Suny Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Kaiser Permanente Oncology/Hematology, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke'S Hospital & Health Network Laboratory, Bethlehem, Pennsylvania
  - Cancer Center Of The Carolinas, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Scott & White Memorial Hospital And Clinic, Temple, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Providence Regional Medical Center Everett, Everett, Washington
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, La Rioja, La Rioja Province
  - Local Institution, Rosario, Santa Fe Province
- Australia (7):
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Ashford, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, East Bentleigh, Victoria
  - Local Institution, Frankston, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Subiaco, Western Australia
- Brazil (5):
  - Local Institution, Brasília, Federal District
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Belo Horizonte - Mg, Minas Gerais
  - Local Institution, Ijuí, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
- Canada (3):
  - Local Institution, Kingston, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Chile (3):
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago
- Colombia (4):
  - Local Institution, Montería, Departamento de Córdoba
  - Local Institution, Bogotá
  - Local Institution, Bucaramanga
  - Local Institution, Medellín
- Czechia (3):
  - Local Institution, Hradec Králové
  - Local Institution, Liberec
  - Local Institution, Prague
- Denmark (2):
  - Local Institution, Herlev
  - Local Institution, København Ø
- France (6):
  - Local Institution, Bordeaux
  - Local Institution, Clermont-Ferrand
  - Local Institution, Marseille
  - Local Institution, Pointe à Pitre
  - Local Institution, Poitiers
  - Local Institution, Villejuif
- Germany (5):
  - Local Institution, Aachen
  - Local Institution, Heidelberg
  - Local Institution, Marktredwitz
  - Local Institution, Munich
  - Local Institution, Wesel
- Local Institution, Athens, Greece
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Gyula
  - Local Institution, Székesfehérvár
- Italy (4):
  - Local Institution, Meldola (FC)
  - Local Institution, Milan
  - Local Institution, Siena
  - Local Institution, Terni
- Mexico (6):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, México, Querétaro
  - Local Institution, San Luis Potosí City, San Luis Potosí
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Sittard-geleen
- Local Institution, Kristiansand, Norway
- Poland (7):
  - Local Institution, Gdansk
  - Local Institution, Kościerzyna
  - Local Institution, Krakow
  - Local Institution, Kutno
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Słupsk
- Va Caribbean Healthcare System, San Juan, Puerto Rico
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Cluj-napoca, Cluj County
  - Local Institution, Timisoara,timis County
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Seville
  - Local Institution, Valencia
- Sweden (3):
  - Local Institution, Stockholm
  - Local Institution, Uppsala
  - Local Institution, Vaxjo
- Turkey (Türkiye) (4):
  - Local Institution, Adana
  - Local Institution, Bornova, Izmir
  - Local Institution, Gaziantep
  - Local Institution, Kocaeli
- United Kingdom (3):
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Guildford, Surrey
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180
- [Derived] Dayyani F, Gallick GE, Logothetis CJ, Corn PG. Novel therapies for metastatic castrate-resistant prostate cancer. J Natl Cancer Inst. 2011 Nov 16;103(22):1665-75. doi: 10.1093/jnci/djr362. Epub 2011 Sep 13. PMID 21917607
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 837 participants enrolled; 602 randomized; 598 treated. Of the 235 not randomized, 189 no longer met criteria, 28 withdrew consent, 2 suffered Adverse Events, 2 were non-compliant, 1 was lost to follow-up, and 13 were removed for other/unspecified reasons. Post-randomization, 4 no longer met criteria and were not treated (3 placebo, 1 ipilimumab)
Groups:
- Placebo: Placebo infusion (normal saline or 5% dextrose) 2mL/kg was administered intravenously (IV) over 90 minutes. Induction dosing occurred on Days 1, 22, 43, and 64 during the Induction phase and every 12 weeks starting at Week 24 during the Maintenance phase until unacceptable toxicity, clinical deterioration, confirmed disease progression, or study closure.
- Ipilimumab: Ipilimumab 10 mg/kg was administered intravenously (IV) over 90 minutes with a normal saline flush at the end. Induction dosing occurred on Days 1, 22, 43, and 64 during the Induction phase and every 12 weeks starting at Week 24 during the Maintenance phase until unacceptable toxicity, clinical deterioration, confirmed disease progression, or study closure.
Period: Overall Study
Arm/Group | Placebo | Ipilimumab
Started | 199 | 399
Completed | 1 | 1
Not Completed | 198 | 398
Not completed — Disease progression | 156 | 197
Not completed — Study drug toxicity | 5 | 114
Not completed — Adverse event unrelated to study drug | 13 | 29
Not completed — Withdrawal by Subject | 10 | 25
Not completed — Death | 2 | 12
Not completed — Maximum clinical benefit | 5 | 5
Not completed — Poor/non-compliance | 0 | 1
Not completed — No longer met study criteria | 0 | 1
Not completed — Other | 7 | 14

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ipilimumab | Total
Number analyzed (Participants) | 202 | 400 | 602
Age, Continuous [Mean (Full Range); unit: years] | 68.6 [42 to 92] | 69.3 [44 to 91] | 69.0 [42 to 92]
Age, Customized [Number; unit: participants]
  < 65 years | 65 | 104 | 169
  >= 65 years | 137 | 296 | 433
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 202 | 400 | 602
Region of Enrollment [Number; unit: participants]
  North America | 79 | 154 | 233
  South America | 25 | 52 | 77
  Europe | 74 | 161 | 235
  Australia | 24 | 33 | 57

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: OS was defined as the time from the date of randomization until the date of death. For participants without documentation of death, OS was censored at the last date the participant was known to be alive.
Time Frame: Randomization until death from any cause, up to April 2015, approximately 57 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ipilimumab
Number analyzed (Participants) | 202 | 400
months | 29.73 [26.12 to 34.17] | 28.65 [24.48 to 32.46]
Statistical Analysis 1: Comparison: Placebo vs Ipilimumab; Test type: Superiority or Other; p = 0.3667, Log Rank; Hazard Ratio (HR) = 1.11, 95.87% CI 2-sided [0.88 to 1.39] — Hazard ratio = ipilimumab over placebo

2. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: Progression-free survival, as determined by the investigator, was defined as the time from randomization to the earliest date of confirmed Prostate-Specific Antigen (PSA) progression, confirmed radiological progression, clinical deterioration, or death.
Time Frame: Randomization until disease progression, up to April 2015, approximately 57 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ipilimumab
Number analyzed (Participants) | 202 | 400
months | 3.81 [2.76 to 4.11] | 5.59 [5.32 to 6.28]
Statistical Analysis 1: Comparison: Placebo vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.55 to 0.80] — HR = ipilimumab over placebo

3. Secondary Outcome: Time to Subsequent Non-hormonal Cytotoxic Therapy
Description: For participants who discontinued treatment or experienced disease progression while on study therapy and then received subsequent non-hormonal cytotoxic therapy, time to subsequent non-hormonal cytotoxic therapy was defined as the time from randomization to the time of initiation of subsequent non-hormonal cytotoxic therapy. Participants who did not receive subsequent non-hormonal cytotoxic therapy were censored on the last known alive date (for participants who have not died) or the date of last follow-up contact at which the participants was known alive (for participants who died).
Time Frame: Randomization until subsequent non-hormonal cytotoxic therapy, up to April 2015, approximately 57 months
Population: All randomized participants who received subsequent non-hormonal cytotoxic therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ipilimumab
Number analyzed (Participants) | 128 | 199
months | 10.91 [8.44 to 14.59] | 18.04 [15.18 to 24.80]
Statistical Analysis 1: Comparison: Placebo vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.65, 95.87% CI 2-sided [0.52 to 0.83] — HR = Ipilimumab over placebo

4. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time from randomization to the time of the earliest date of any of the following 4 events: 1) an increase in average daily worst pain intensity of >= 2 points from baseline according to the Brief Pain Inventory - Short Form (BPI-SF), maintained over 2 consecutive time periods. 2) initiation of opioid analgesic (excluding codeine or dextropropoxyphene). 3) initiation of palliative radiotherapy for prostate cancer. 4) increase in mean Analgesic Score (AS) of >= 25% from baseline (for participants with baseline AS > 10) or increase in mean AS >= 10 points from baseline (for participants with baseline AS <= 10).
  Participants who did not experience any of these events were censored on the earliest date among the latest BPI-SF completion date with non-missing worst pain assessment and last evaluable disease assessment date as defined in the PFS censoring mechanism.
Time Frame: Randomization until pain progression, up to April 2015, approximately 57 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ipilimumab
Number analyzed (Participants) | 202 | 400
months | 16.62 [11.53 to NA] — Upper bounds were not estimable due to censoring | 21.68 [19.22 to NA] — Upper bounds were not estimable due to censoring
Statistical Analysis 1: Comparison: Placebo vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.98, 95.87% CI 2-sided [0.71 to 1.35] — HR = Ipilimumab over placebo

5. Secondary Outcome: Number of Participants Who Died or Had Adverse Events (AEs), Serious Adverse Events (SAEs), Immune-related AEs (irAEs), or Immune-mediated Adverse Reactions (imARs)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. irAE=AEs consistent with an immune mediated mechanism. imAR=AEs of special interest that were adjudicated as imAR by investigator. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Events were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Day 1 of study therapy to last dose plus 70 days
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Placebo | Ipilimumab
Number analyzed (Participants) | 199 | 399
participants
  AE (grade 3-4) | 59 | 223
  Drug-related AE (any grade) | 98 | 325
  Drug-related AE (grade 3-4) | 11 | 158
  SAE (any grade) | 53 | 213
  SAE (grade 3-4) | 39 | 153
  AE leading to DC (any grade) | 20 | 139
  AE leading to DC (grade 3-4) | 14 | 103
  irAE (any grade) | 57 | 309
  irAE (grade 3-4) | 3 | 125
  imAR (grade >= 2) | 14 | 273
  Deaths | 130 | 259

6. Secondary Outcome: Number of Treated Participants With Grade 3 or 4 Clinical Laboratory Abnormalities
Description: NCI CTC, Version 3 used to assess parameters. LLN=lower limit of normal. ULN=upper limit of normal. CTC criteria:
  White blood cells (WBC): Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L. Absolute neutrophil count (ANC): Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L.
  Platelet count: Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Hemoglobin: Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Absolute Lymphocyte Count (ALC): Gr 3: 0.2 - <0.5*10^9/L, Gr 4: <0.2*10^9/L.
  Lipase: Gr 3:> 2.0 - 5.0 * ULN; Gr 4: > 5.0 X ULN. Amylase: Gr 3: > 2.0 - 5.0 * ULN; Gr 4: > 5.0 * ULN. Alanine Aminotransferase (ALT) Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Aspartate Aminotransferase (AST): Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Bilirubin: Gr 3: > 3.0 - 10.0 * ULN; Gr 4: > 10.0 * ULN. Alkaline Phosphatase: Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Creatinine: Gr 3: > 3.0-6.0 * ULN, Gr 4: >6.0 * ULN.
Time Frame: Randomization up to April 2015, approximately 57 months
Population: All treated participants with on-study laboratory results
Measure: Number; unit: participants
Arm/Group | Placebo | Ipilimumab
Number analyzed (Participants) | 198 | 386
participants
  WBC (n=195;383) | 0 | 3
  ANC (n=195;383) | 0 | 2
  Platelet count (n=194;381) | 0 | 2
  Hemoglobin (n=195;383) | 2 | 5
  ALC (n=195;383) | 4 | 12
  Lipase (n=196;382) | 4 | 27
  Amylase (n=198;385) | 2 | 9
  ALT (n=198;386) | 1 | 16
  AST (n=196;383) | 1 | 18
  Total Bilirubin (n=198;386) | 0 | 4
  Alkaline phosphatase (n=196;383) | 11 | 18
  Creatinine (n=9;23) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of study therapy to last dose plus 70 days
Groups:
- 10 MG/KG IPILIMUMAB: Ipilimumab 10 mg/kg was administered intravenously (IV) over 90 minutes with a normal saline flush at the end. Induction dosing occurred on Days 1, 22, 43, and 64 during the Induction phase and every 12 weeks starting at Week 24 during the Maintenance phase until unacceptable toxicity, clinical deterioration, confirmed disease progression, or study closure.
Arm/Group | PLACEBO | 10 MG/KG IPILIMUMAB
Serious Adverse Events (participants affected / at risk) | 53/199 | 213/399
Other Adverse Events (participants affected / at risk) | 166/199 | 361/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=199) | 10 MG/KG IPILIMUMAB (N=399)
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abscess (Infections and infestations) | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Death (General disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 3
Depressed mood (Psychiatric disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 47
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 2
Obstructive uropathy (Renal and urinary disorders) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 13
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 6 | 2
Vomiting (Gastrointestinal disorders) | 1 | 6
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 29
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Febrile infection (Infections and infestations) | 0 | 1
Fibrosis (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Peripheral swelling (General disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Renal failure (Renal and urinary disorders) | 1 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Adrenal insufficiency (Endocrine disorders) | 0 | 6
Alanine aminotransferase increased (Investigations) | 0 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 8
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 3
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 12
Infected skin ulcer (Infections and infestations) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Malaise (General disorders) | 0 | 3
Motor dysfunction (Nervous system disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 6
Atrial flutter (Cardiac disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Bandaemia (Blood and lymphatic system disorders) | 0 | 2
Bone marrow disorder (Blood and lymphatic system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 14
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 4
Ileus paralytic (Gastrointestinal disorders) | 0 | 2
Impaired healing (General disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 12
Melaena (Gastrointestinal disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 14
Spinal cord compression (Nervous system disorders) | 2 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 5
Asthenia (General disorders) | 0 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 2 | 11
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 4
Headache (Nervous system disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 4
Hypothyroidism (Endocrine disorders) | 0 | 2
IVth nerve paresis (Nervous system disorders) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Meningitis aseptic (Infections and infestations) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 8
VIIth nerve paralysis (Nervous system disorders) | 0 | 2
Weight decreased (Investigations) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Haemorrhagic infarction (Vascular disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 2
Megacolon (Gastrointestinal disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Multi-organ failure (General disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sudden death (General disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
Transaminases increased (Investigations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 2
Cluster headache (Nervous system disorders) | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 2
Drug dependence (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 1
Embolism (Vascular disorders) | 0 | 1
Endocrine disorder (Endocrine disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Eye disorder (Eye disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Mononeuropathy (Nervous system disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myasthenia gravis crisis (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 10
Pain (General disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 3
Cellulitis (Infections and infestations) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Infection (Infections and infestations) | 0 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pyelonephritis (Infections and infestations) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Secondary hypothyroidism (Endocrine disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Urogenital disorder (Renal and urinary disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=199) | 10 MG/KG IPILIMUMAB (N=399)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 21
Diarrhoea (Gastrointestinal disorders) | 48 | 190
Pollakiuria (Renal and urinary disorders) | 10 | 16
Urinary tract infection (Infections and infestations) | 15 | 31
Vomiting (Gastrointestinal disorders) | 18 | 75
Anaemia (Blood and lymphatic system disorders) | 12 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 51
Abdominal pain (Gastrointestinal disorders) | 13 | 50
Alanine aminotransferase increased (Investigations) | 1 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 69
Hot flush (Vascular disorders) | 11 | 15
Hypertension (Vascular disorders) | 7 | 24
Aspartate aminotransferase increased (Investigations) | 2 | 27
Dehydration (Metabolism and nutrition disorders) | 6 | 31
Pyrexia (General disorders) | 18 | 63
Asthenia (General disorders) | 20 | 61
Fatigue (General disorders) | 55 | 144
Haematuria (Renal and urinary disorders) | 11 | 13
Headache (Nervous system disorders) | 24 | 73
Hypotension (Vascular disorders) | 6 | 21
Hypothyroidism (Endocrine disorders) | 0 | 25
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 45
Weight decreased (Investigations) | 17 | 61
Constipation (Gastrointestinal disorders) | 37 | 84
Decreased appetite (Metabolism and nutrition disorders) | 30 | 114
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 25
Oedema peripheral (General disorders) | 9 | 44
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 123
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 45
Dizziness (Nervous system disorders) | 17 | 39
Insomnia (Psychiatric disorders) | 9 | 38
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 27 | 41
Nausea (Gastrointestinal disorders) | 36 | 115
Pain (General disorders) | 17 | 25
Vision blurred (Eye disorders) | 1 | 21
Dysgeusia (Nervous system disorders) | 6 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 33
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 24
Rash (Skin and subcutaneous tissue disorders) | 22 | 145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.